CLINICAL TRIAL: NCT04970069
Title: The Effect of Preoperative Education on Postoperative Opioid Consumption
Brief Title: Preoperative Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 21-626
Record Dates: First submitted 2021-07-16; First posted 2021-07-21 (Actual); Results first posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Analgesic education (Active Comparator)
  Interventions: Other: Video on analgesic education
- General perioperative education (Placebo Comparator)
  Interventions: Other: Video on general perioperative education

INTERVENTIONS:
Other: Video on analgesic education — A four minute video informing the patient about opioids.
  Arms: Analgesic education
Other: Video on general perioperative education — A four minute video informing the patient about general perioperative process.
  Arms: General perioperative education

SUMMARY:
The investigators will evaluate the effect of preoperative education on postoperative opioid.

DETAILED DESCRIPTION:
The investigators propose a randomized trial to be performed at the Cleveland Clinic. Patients will be assigned to: 1) an educational video focused on postoperative analgesia modalities, opioids, and realistic pain expectations (analgesic education); or, 2) an educational video focused on other aspects of the perioperative experience.

ELIGIBILITY:
Inclusion Criteria:

* Modified informed consent
* Adults ≥18 years
* American Society of Anaesthesiologists physical status 1-4
* Scheduled for hip arthroplasty, laparoscopy assisted colorectal surgery
* Personal visit the PACE clinic
* Anticipated overnight postoperative hospitalization
* Reasonable English fluency

Exclusion Criteria:

* Opioid use for more than 30 consecutive days within three preoperative months, at a daily dose of 15 mg or more of morphine or equivalent
* Regional block or epidural analgesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1057 (Actual)
Dates: Start 2021-07-25 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alparslan Turan, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Analgesic Education | General Perioperative Education
Started | 527 | 530
Completed | 483 | 474
Not Completed | 44 | 56

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Analgesic Education | General Perioperative Education | Total
Number analyzed (Participants) | 527 | 530 | 1057
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Excludes patients not analyzed due to surgical cancellations/reschedule, and randomization errors.
  years
    number analyzed (Participants) | 483 | 474 | 957
    (all) | 60 (15) | 60 (15) | 60 (15)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Excludes patients not analyzed due to surgical cancellations/reschedule, and randomization errors.
  Participants
    number analyzed (Participants) | 483 | 474 | 957
    Female | 193 | 198 | 391
    Male | 290 | 276 | 566
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Excludes patients not analyzed due to surgical cancellations/reschedule, and randomization errors.
  Participants
    Black: number analyzed (Participants) | 483 | 474 | 957
    Black | 67 | 55 | 122
    White: number analyzed (Participants) | 483 | 474 | 957
    White | 388 | 393 | 781
    Other: number analyzed (Participants) | 483 | 474 | 957
    Other | 28 | 26 | 54
Region of Enrollment [Number; unit: participants]
  United States | 527 | 530 | 1057
History of chronic pain [Count of Participants; unit: Participants] — Population: Excludes patients not analyzed due to surgical cancellations/reschedule, and randomization errors.
  Participants
    number analyzed (Participants) | 483 | 474 | 957
    (all) | 15 | 20 | 35
Type of surgery [Count of Participants; unit: Participants] — Population: Excludes patients not analyzed due to surgical cancellations/reschedule, and randomization errors.
  Participants
    Laparoscopic colorectal: number analyzed (Participants) | 483 | 474 | 957
    Laparoscopic colorectal | 24 | 21 | 45
    Orthopedic: number analyzed (Participants) | 483 | 474 | 957
    Orthopedic | 51 | 63 | 114
    Laparoscopic abdominal: number analyzed (Participants) | 483 | 474 | 957
    Laparoscopic abdominal | 408 | 390 | 798

OUTCOME MEASURES:

1. Primary Outcome: Opioid Consumption
Description: Opioid consumption (morphine milligrams equivalent) during the initial 72 hours after surgery.
Time Frame: 72 hours after surgery
Population: Modified intention to treat analysis population
Measure: Median (Inter-Quartile Range); unit: Morphine milligrams equivalent
Arm/Group | Analgesic Education | General Perioperative Education
Number analyzed (Participants) | 483 | 474
Morphine milligrams equivalent | 23 [13 to 42] | 26 [10 to 45]
Statistical Analysis 1: Comparison: Analgesic Education vs General Perioperative Education; Multiple imputation by chained equations (MICE) was used for imputing missing outcomes and covariates; Test type: Superiority; p = 0.890, Regression, Linear; Ratio of geometric means = 1.01, 95% CI 2-sided [0.86 to 1.18] — The numerator and denominator for the ratio of geometric means are analgesic education and general preoperative education respectively

2. Secondary Outcome: Time-weighted Average Pain Scores
Description: Time-weighted average of pain scores obtained from electronic medical records. Pain scores were measured using the numeric rating scale ranging from 0-10, with 0 indicating the lowest pain (better) and 10 the highest pain (worse). Pain scores were recorded approximately every 15 minutes in the post-anesthesia care unit and then every 4 hours in the ward.
Time Frame: 72 hours after surgery, or until discharge, whichever was earlier
Population: Modified intention to treat population
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Analgesic Education | General Perioperative Education
Number analyzed (Participants) | 483 | 474
score on a scale | 4 [3 to 5] | 4 [3 to 5]
Statistical Analysis 1: Comparison: Analgesic Education vs General Perioperative Education; Test type: Superiority; p = 0.617, Regression, Linear; Median Difference (Final Values) = -0.1, 95% CI 2-sided [-0.3 to 0.2]

3. Secondary Outcome: Satisfaction With Post Operative Pain Management
Description: Patient satisfaction measured using Likert scale 0-10 with 0 meaning not satisfied and 10 meaning completely satisfied.
Time Frame: 3 days after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Analgesic Education | General Perioperative Education
Number analyzed (Participants) | 483 | 474
score on a scale | 9 [8 to 10] | 10 [8 to 10]
Statistical Analysis 1: Comparison: Analgesic Education vs General Perioperative Education; Test type: Superiority; p = 0.611, Regression, Linear; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.3 to 0.2]

ADVERSE EVENTS:
Time Frame: 72 hours after surgery or until discharge, whichever was earlier.
Arm/Group | Analgesic Education | General Perioperative Education
All-Cause Mortality (participants affected / at risk) | 0/483 | 2/474
Serious Adverse Events (participants affected / at risk) | 0/483 | 0/474
Other Adverse Events (participants affected / at risk) | 181/483 | 176/474
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Analgesic Education (N=483) | General Perioperative Education (N=474)
Ileus (Gastrointestinal disorders) | 27 | 23
Nausea and vomiting (Gastrointestinal disorders) | 22 | 28
Urinary catheterization (Renal and urinary disorders) | 15 | 26
Anti-emetic use (Gastrointestinal disorders) | 156 | 155

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-04): https://cdn.clinicaltrials.gov/large-docs/69/NCT04970069/Prot_SAP_000.pdf